CLINICAL TRIAL: NCT00272987
Title: A Randomized, Double Blind, Placebo-Controlled, Multicenter, Phase III Study Comparing the Activity of Paclitaxel Plus Trastuzumab Plus Lapatinib to Paclitaxel Plus Trastuzumab Plus Placebo in Women With ErbB2 Overexpressing Metastatic Breast Cancer
Brief Title: ErbB2 Over-expressing Metastatic Breast Cancer Study Using Paclitaxel, Trastuzumab, and Lapatinib
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment was closed after the open label stage due to poor recruitment rate (randomized stage never opened).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EGF104383; 2005-003432-22 (EudraCT Number); CLAP016A2301 (Other: Novartis)
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Neoplasms, Breast
Keywords: trastuzumab; ErbB2; paclitaxel; Herceptin; Taxol; ErbB1; metastatic breast cancer; Stage IV breast cancer; lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants received: paclitaxel 80mg/m2 IV weekly for 3 weeks of a 4 week cycle plus trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly plus lapatinib 1000 mg PO daily
  Interventions: Drug: lapatinib; Drug: paclitaxel; Drug: trastuzumab
- Cohort 2 (Experimental): Participants received paclitaxel 70mg/m2 IV weekly for 3 weeks of a 4 week cycle plus trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly plus lapatinib 1000 mg PO daily.
  Interventions: Drug: lapatinib; Drug: paclitaxel; Drug: trastuzumab
- Cohort 3 (Experimental): Participants in this arm received 80mg/m2 IV weekly for 3 weeks of a 4 week cycle plus trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly plus lapatinib 750 mg PO
  Interventions: Drug: lapatinib; Drug: paclitaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: lapatinib — (GW572016) 1000 mg QD
Drug: paclitaxel — 80 mg/m2 IV weekly for three weeks
Drug: trastuzumab — 4 mg/kg loading dose and 2 mg/kg weekly IV

SUMMARY:
This study was originally designed as a Phase III randomized, double blind, placebo controlled study to assess the safety and tolerability, and efficacy of paclitaxel plus trastuzumab plus lapatinib compared with paclitaxel plus trastuzumab plus placebo in women with ErbB2 overexpressing metastatic breast cancer. The planned study was a two stage design with an initial open-label safety stage to be conducted in approximately 65 subjects followed by a randomized phase conducted in a further 700 subjects. The open-label part of the study sequentially enrolled three cohorts with patients receiving a different dose combination of paclitaxel, trastuzumab and lapatinib. Following poor recruitment rate in the open label stage, the randomized stage of the study was terminated, thus no subjects were enrolled into the randomization stage.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate and compare time to progression (TTP). The Primary objective for open label phase was to determine the safety and tolerability of lapatinib when administered in combination with both paclitaxel and trastuzumab. The study first enrolled an open label safety cohort of 20 patients to assess the tolerability of the triplet combination. This was a 1 arm, 3 cohort study stage.

Open-label Phase: Patients were sequentially enrolled into three cohorts and received an open-label combination of paclitaxel, trastuzumab and lapatinib: Cohort 1 received paclitaxel 80mg/m2 IV weekly for 3 weeks of a 4 week cycle, trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly, and lapatinib 1000 mg PO daily. Cohort 2 received paclitaxel 70mg/m2 IV weekly for 3 weeks of a 4 week cycle, trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly, and lapatinib 1000 mg PO daily. Cohort 3 paclitaxel 80mg/m2 IV weekly for 3 weeks of a 4 week cycle, trastuzumab 4 mg/kg IV loading dose and 2 mg/kg IV weekly, and lapatinib 750 mg PO daily.

Randomized Phase: was terminated following the poor recruitment rate in the open-label safety stage. No subjects were enrolled into the randomization stage.

In summary, at approximately 3.5 years the primary analysis which included demographics, efficacy and safety were conducted; at approximately 7 years protocol amendment 7 cancelled collection of efficacy endpoints, and only key safety endpoints were to be collected; the final analysis was performed at approximately 14 years.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed invasive breast cancer with stage IV disease
* If trastuzumab was administered in the adjuvant setting, >12 months must have elapsed since discontinuation of trastuzumab therapy
* If a taxane was administered in the neoadjuvant or adjuvant setting, progression must have occurred ≥12 months after completion of this treatment
* Had tumors that overexpress ErbB2 defined as either: 3+ by IHC OR c-erbB2 gene amplification by FISH OR 0, 1+, 2+ by IHC and c-erbB2 gene amplification by FISH.
* Patients must have tumor tissue available for central testing, and must have Measurable lesion(s) according to RECIST
* Subjects must be females of at least 18 years Non-childbearing potential or Childbearing potential but using adequate contraception
* Radiotherapy to a limited area other than the sole site of measurable and assessable disease is allowed; however, patients must have completed treatment and recovered from all acute treatment-related toxicities prior to administration of the first dose of study medication
* Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of randomized therapy. Prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
* For those patients whose disease is estrogen receptor positive+ and/or progesterone receptor + one the following criteria should be met: Patients with visceral disease that requires chemotherapy (eg., patients with liver or lung metastases) or Rapidly progressing/life threatening disease, as determined by the investigator or Patients who received hormonal therapy and are no longer benefiting from this therapy;
* Able to swallow and retain oral medication
* Cardiac ejection fraction within institutional range of normal
* Patient must have adequate organ function

Exclusion criteria:

* Pregnant or lactating females;
* Received prior chemotherapy, immunotherapy, biologic therapy, or anti-ErbB1/ErbB2 therapy for metastatic disease, prior hormonal therapy is permitted but must be discontinued a minimum of 7 days prior to randomization;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Patients with ulcerative colitis are also excluded;
* History of other malignancy; however, patients who have been disease-free for five years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible;
* Concurrent disease or condition that would make the patient inappropriate for study participation, or any serious medical disorder that would interfere with the patient's safety;
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment;
* Peripheral neuropathy of Grade 2 or greater;
* Active or uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* Known history of uncontrolled or symptomatic angina, arrhythmias, conduction abnormalities or congestive heart failure;
* Known history or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis;
* Concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy);
* Concurrent treatment with an investigational agent or participation in another clinical trial;
* Concurrent treatment with any medication on the prohibited medications list.
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of treatment. Hormonal therapy needs to be discontinued at least 7 days before the first dose of treatment.
* Prior therapy with an ErbB2 inhibitor, other than trastuzumab in the adjuvant setting;
* A known immediate or delayed hypersensitivity reaction to drugs chemically related to lapatinib or excipients;
* A known immediate or delayed hypersensitivity reaction to drugs chemically related to paclitaxel or excipients;
* A known immediate or delayed hypersensitivity reaction to drugs chemically related to trastuzumab or excipients;
* Non compliance with any of the screening procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-12-13 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (13):
  - Novartis Investigative Site, Roswell, Georgia
  - Novartis Investigative Site, Joliet, Illinois
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Middletown, Ohio
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Belgium (2):
  - Novartis Investigative Site, Arlon
  - Novartis Investigative Site, Liège

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Esteva FJ, Franco SX, Hagan MK, Brewster AM, Somer RA, Williams W, Florance AM, Turner S, Stein S, Perez A. An open-label safety study of lapatinib plus trastuzumab plus paclitaxel in first-line HER2-positive metastatic breast cancer. Oncologist. 2013 Jun;18(6):661-6. doi: 10.1634/theoncologist.2012-0129. Epub 2013 May 22. PMID 23697602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female participants (par.) with histologically confirmed invasive breast cancer (Stage IV disease) whose tumors overexpressed the ErbB2 protein, documented by either Immunohistochemistry (IHC) or fluorescence in situ hybridisation (FISH), were eligible for inclusion in this study.
Pre-assignment Details: Participants who met inclusion criteria were sequentially enrolled into three cohorts and received the open-label triple combination of paclitaxel, trastuzumab and lapatinib. The planned randomized phase of the study was terminated following the poor recruitment rate in the Open-label Phase.
Groups:
- Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg: Participants received an intravenous (IV) infusion of paclitaxel 80 milligrams per meter squared (mg/m^2) over 60 minutes weekly for 3 weeks of a 4-week cycle plus an IV infusion of trastuzumab 4 mg per kilogram (mg/kg) loading dose and 2 mg/kg weekly plus a daily dose of 4 tablets of lapatinib (total daily dose 1000 mg) at approximately the same time every day, either 1 hour (or more) before a meal or 1 hour (or more) after a meal.
- Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg: Participants received an IV infusion of paclitaxel 70 mg/m^2 over 60 minutes weekly for 3 weeks of a 4-week cycle plus an IV infusion of trastuzumab 4 mg/kg loading dose and 2 mg/kg weekly plus a daily dose of 4 tablets of lapatinib (total daily dose 1000 mg) at approximately the same time every day, either 1 hour (or more) before a meal or 1 hour (or more) after a meal. The paclitaxel dose was systematically increased to 80 mg/m^2 after 2 cycles if 70 mg/m^2 was tolerated.
- Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg: Participants received an IV infusion of paclitaxel 80 mg/m^2 over 60 minutes weekly for 3 weeks of a 4-week cycle plus an IV infusion of trastuzumab 4 mg/kg loading dose and 2 mg/kg weekly plus a daily dose of 3 tablets of lapatinib (total daily dose 750 mg) at approximately the same time every day, either 1 hour (or more) before a meal or 1 hour (or more) after a meal. The lapatinib dose was systematically increased to 1000 mg after 2 cycles if the 750 mg dose was tolerated.
Period: Overall Study
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Started | 29 | 14 | 20
Completed | 20 | 10 | 9
Not Completed | 9 | 4 | 11
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Sponsor Terminated study | 0 | 1 | 1
Not completed — Disease progression | 1 | 1 | 2
Not completed — Non-compliant- study visits, trtmnts, req. surgery | 2 | 1 | 4
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg | Total
Number analyzed (Participants) | 29 | 14 | 20 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (11.08) | 56.1 (11.92) | 52.2 (13.00) | 52.7 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 14 | 20 | 63
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 7 | 2 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 22 | 11 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Extent of Exposure to Lapatinib, Trastuzumab and Paclitaxel by Mean/Standard Deviation
Description: Extent of exposure is defined as the duration of the treatment administered during the study. The mean duration of exposure to lapatinib, trastuzumab and paclitaxel is calculated as the number of weeks between the start and end of treatment.
Time Frame: From the date of the first dose of the investigational product to end of study, up to approx. 14 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Weeks
  Lapatinib | 70.9 (115.44) | 93.1 (147.92) | 82.5 (135.79)
  Trastuzumab | 60.7 (72.07) | 72.2 (88.66) | 62.3 (75.52)
  Paclitaxel | 26.9 (16.88) | 29.4 (23.00) | 23.8 (14.87)

2. Primary Outcome: Extent of Exposure to Lapatinib, Trastuzumab and Paclitaxel by Median/Min-Max
Description: as for outcome 1
Time Frame: From the date of the first dose of the investigational product to end of study, up to approx. 14 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Weeks
  Lapatinib | 33.0 [3 to 615] | 38.5 [2 to 547] | 32.5 [1 to 574]
  Trastuzumab | 33.0 [2 to 343] | 37.0 [2 to 271] | 31.5 [1 to 245]
  Paclitaxel | 22.0 [2 to 86] | 23.5 [2 to 94] | 22.0 [1 to 63]

3. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Refer to the general AE/SAE module for a list of non-serious AEs and SAEs.
Time Frame: From the date of the first dose of investigational product until 30 days after the last dose of investigational product, up to approx. 14 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants
  Any AEs | 29 | 14 | 20
  Any SAEs | 14 | 6 | 5

4. Primary Outcome: Number of Participants Who Died Due to Any Cause
Description: Number of participants who died due to any cause throughout the study including off-treatment deaths (on-treatment deaths are reported for the All-Cause Mortality in the AE section).
Time Frame: From the date of the first dose of investigational product until last patient last visit, up to approximately 14 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants | 12 | 2 | 1

5. Primary Outcome: Number of Events of Diarrhea With the Indicated Characteristics
Description: Events of diarrhea are characterized as serious, related to investigational product, leading to withdrawal from the study and fatal. Participants could have been counted in more than one category.
Time Frame: From the date of the first dose of investigational product until 30 days after the last dose of investigational product, up to approx. 3.5 years
Population: Safety Population. Only the participants with at least one event of diarrhea were analyzed.
Measure: Number; unit: Events of diarrhea
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 28 | 13 | 13
Events of diarrhea
  Any Event | 358 | 90 | 37
  Serious | 4 | 0 | 0
  Related to investigational product | 347 | 75 | 26
  Leading to withdrawal from study | 2 | 1 | 1
  Fatal | 0 | 0 | 0

6. Primary Outcome: Number of Events of Rash With the Indicated Characteristics
Description: Events of rash are characterized as serious, related to investigational product, leading to withdrawal from the study and fatal. Participants could have been counted in more than one category.
Time Frame: as for outcome 5
Population: Safety Population. Only the participants with at least one event of rash were analyzed.
Measure: Number; unit: Events of rash
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 24 | 8 | 15
Events of rash
  Any Event | 69 | 23 | 20
  Serious | 2 | 0 | 0
  Related to investigational product | 55 | 12 | 7
  Leading to withdrawal from study | 3 | 0 | 0
  Fatal | 0 | 0 | 0

7. Primary Outcome: Number of Participants With the Maximum Toxicity Grade for the Indicated Clinical Hematology Parameters
Description: Blood samples for clinical laboratory evaluation were taken at Baseline prior to the administration of investigational product and thereafter at each scheduled visit. Haematology parameters included haemoglobin, total white blood cell count (WBC), neutrophils, lymphocytes and platelets. Hematology data was summarized by the National Cancer Institute's Common toxicity criteria for adverse events (NCI CTCAE) toxicity grade (Version 3.0). Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling; Grade 5, death.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants
  Haemaglobin, Grade 1 | 19 | 11 | 11
  Haemaglobin, Grade 2 | 7 | 1 | 6
  Haemaglobin, Grade 3 | 2 | 0 | 1
  Haemaglobin, Grade 4 | 1 | 0 | 0
  Platelets, Grade 1 | 3 | 0 | 0
  Platelets, Grade 2 | 1 | 0 | 0
  Platelets, Grade 3 | 0 | 0 | 0
  Platelets, Grade 4 | 1 | 0 | 0
  Total WBC, Grade 1 | 10 | 6 | 7
  Total WBC, Grade 2 | 8 | 4 | 2
  Total WBC, Grade 3 | 3 | 1 | 4
  Total WBC, Grade 4 | 1 | 0 | 0
  Neutrophils, Grade 1 | 7 | 2 | 5
  Neutrophils, Grade 2 | 7 | 4 | 4
  Neutrophils, Grade 3 | 3 | 1 | 5
  Neutrophils, Grade 4 | 3 | 0 | 0
  Lymphocytes, Grade 1 | 5 | 3 | 7
  Lymphocytes, Grade 2 | 10 | 4 | 4
  Lymphocytes, Grade 3 | 5 | 3 | 1
  Lymphocytes, Grade 4 | 1 | 0 | 1

8. Primary Outcome: Number of Participants With the Maximum Toxicity Grade for the Indicated Clinical Chemistry Parameters
Description: Blood samples for clinical laboratory evaluation were taken at Baseline prior to the administration of investigational product and thereafter at each scheduled visit. Clinical chemistry parameters included values > upper limit of normal (ULN)=Hyper; values < lower limit of normal (LLN)=Hypo of sodium (Hypernatraemia and Hyponatraemia), potassium (Hyperkalaemia and Hypokalaemia), calcium (Hypercalcaemia and Hypocalcaemia), glucose (Hyperglycaemia and Hyperglycaemia), creatinine (if >2 milligram per deciliter [mg/dL]), aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phophatase, total bilirubin (if available bilirubin fractionation is recommended if the total bilirubin is > twice of ULN), and albumin. Clinical chemistry data was summarized by National Cancer Institute's Common toxicity criteria for adverse events (NCI CTCAE) toxicity grade (Version 3.0). Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling; Grade 5, death.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants
  Hypernatraemia, Grade 1 | 0 | 1 | 1
  Hypernatraemia, Grade 2 | 1 | 0 | 0
  Hypernatraemia, Grade 3 | 0 | 0 | 0
  Hypernatraemia, Grade 4 | 0 | 0 | 0
  Hyponatraemia, Grade 1 | 8 | 1 | 1
  Hyponatraemia, Grade 2 | 0 | 0 | 0
  Hyponatraemia, Grade 3 | 0 | 1 | 0
  Hyponatraemia, Grade 4 | 0 | 0 | 0
  Hyperkalaemia, Grade 1 | 2 | 0 | 0
  Hyperkalaemia, Grade 2 | 2 | 1 | 1
  Hyperkalaemia, Grade 3 | 0 | 0 | 0
  Hyperkalaemia, Grade 4 | 1 | 0 | 1
  Hypokalaemia, Grade 1 | 11 | 6 | 6
  Hypokalaemia, Grade 2 | 0 | 0 | 0
  Hypokalaemia, Grade 3 | 6 | 2 | 0
  Hypokalaemia, Grade 4 | 0 | 0 | 0
  Hypercalcaemia, Grade 1: number analyzed (Participants) | 29 | 14 | 19
  Hypercalcaemia, Grade 1 | 1 | 0 | 0
  Hypercalcaemia, Grade 2: number analyzed (Participants) | 29 | 14 | 19
  Hypercalcaemia, Grade 2 | 0 | 0 | 0
  Hypercalcaemia, Grade 3: number analyzed (Participants) | 29 | 14 | 19
  Hypercalcaemia, Grade 3 | 0 | 0 | 0
  Hypercalcaemia, Grade 4: number analyzed (Participants) | 29 | 14 | 19
  Hypercalcaemia, Grade 4 | 0 | 0 | 0
  Hypocalcaemia, Grade 1: number analyzed (Participants) | 29 | 14 | 19
  Hypocalcaemia, Grade 1 | 10 | 3 | 4
  Hypocalcaemia, Grade 2: number analyzed (Participants) | 29 | 14 | 19
  Hypocalcaemia, Grade 2 | 7 | 2 | 3
  Hypocalcaemia, Grade 3: number analyzed (Participants) | 29 | 14 | 19
  Hypocalcaemia, Grade 3 | 3 | 0 | 1
  Hypocalcaemia, Grade 4: number analyzed (Participants) | 29 | 14 | 19
  Hypocalcaemia, Grade 4 | 0 | 0 | 0
  Hyperglycaemia, Grade 1: number analyzed (Participants) | 29 | 14 | 19
  Hyperglycaemia, Grade 1 | 15 | 9 | 6
  Hyperglycaemia, Grade 2: number analyzed (Participants) | 29 | 14 | 19
  Hyperglycaemia, Grade 2 | 3 | 3 | 2
  Hyperglycaemia, Grade 3: number analyzed (Participants) | 29 | 14 | 19
  Hyperglycaemia, Grade 3 | 5 | 0 | 2
  Hyperglycaemia, Grade 4: number analyzed (Participants) | 29 | 14 | 19
  Hyperglycaemia, Grade 4 | 0 | 0 | 0
  Hypoglycemia, Grade 1: number analyzed (Participants) | 29 | 14 | 19
  Hypoglycemia, Grade 1 | 5 | 2 | 2
  Hypoglycemia, Grade 2: number analyzed (Participants) | 29 | 14 | 19
  Hypoglycemia, Grade 2 | 0 | 1 | 1
  Hypoglycemia, Grade 3: number analyzed (Participants) | 29 | 14 | 19
  Hypoglycemia, Grade 3 | 0 | 0 | 0
  Hypoglycemia, Grade 4: number analyzed (Participants) | 29 | 14 | 19
  Hypoglycemia, Grade 4 | 0 | 0 | 0
  Albumin, Grade 1: number analyzed (Participants) | 29 | 14 | 18
  Albumin, Grade 1 | 5 | 3 | 1
  Albumin, Grade 2: number analyzed (Participants) | 29 | 14 | 18
  Albumin, Grade 2 | 3 | 0 | 0
  Albumin, Grade 3: number analyzed (Participants) | 29 | 14 | 18
  Albumin, Grade 3 | 1 | 0 | 0
  Albumin, Grade 4: number analyzed (Participants) | 29 | 14 | 18
  Albumin, Grade 4 | 0 | 0 | 0
  Total Bilirubin, Grade 1 | 2 | 1 | 3
  Total Bilirubin, Grade 2 | 2 | 2 | 1
  Total Bilirubin, Grade 3 | 1 | 1 | 0
  Total Bilirubin, Grade 4 | 0 | 0 | 0
  Creatinine, Grade 1 | 2 | 0 | 0
  Creatinine, Grade 2 | 2 | 0 | 0
  Creatinine, Grade 3 | 1 | 0 | 0
  Creatinine, Grade 4 | 0 | 0 | 0
  Alkaline Phophatase, Grade 1 | 14 | 3 | 5
  Alkaline Phophatase, Grade 2 | 2 | 0 | 0
  Alkaline Phophatase, Grade 3 | 2 | 0 | 0
  Alkaline Phophatase, Grade 4 | 0 | 0 | 0
  ALT, Grade 1 | 7 | 1 | 3
  ALT, Grade 2 | 3 | 3 | 2
  ALT, Grade 3 | 0 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 0
  AST, Grade 1 | 6 | 3 | 6
  AST, Grade 2 | 1 | 1 | 0
  AST, Grade 3 | 1 | 1 | 0
  AST, Grade 4 | 0 | 0 | 0

9. Primary Outcome: Number of Events of Hepatotoxicity With the Indicated Characteristics
Description: Events of hepatotoxicity are characterized as serious, related to investigational product, leading to withdrawal from the study and fatal. Participants could have been counted in more than one category.
Time Frame: as for outcome 5
Population: Safety Population. Only the participants with at least one of event of hepatotoxicity were analyzed.
Measure: Number; unit: Events of hepatotoxicity
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 6 | 0 | 2
Events of hepatotoxicity
  Any Event | 6 |  | 2
  Serious | 0 |  | 0
  Related to investigational product | 5 |  | 0
  Leading to withdrawal from study | 0 |  | 0
  Fatal | 0 |  | 0

10. Primary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at the Indicated Time Points
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Baseline and every 4 weeks thereafter up to withdrawal/study completion and at the 30 day follow-up visit. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
  Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Millimeter of mercury (mmHg)
  SBP, Week 4: number analyzed (Participants) | 28 | 12 | 18
  SBP, Week 4 | 0.5 (16.29) | -7.2 (20.70) | -3.9 (22.76)
  SBP, Week 8: number analyzed (Participants) | 27 | 13 | 17
  SBP, Week 8 | 4.6 (12.35) | -8.6 (22.25) | -2.7 (24.73)
  SBP, Week 12: number analyzed (Participants) | 24 | 12 | 16
  SBP, Week 12 | 3.2 (18.46) | -6.9 (17.09) | -9.3 (23.54)
  SBP, Week 16: number analyzed (Participants) | 23 | 11 | 15
  SBP, Week 16 | 0.8 (18.10) | -6.6 (15.26) | -7.9 (24.43)
  SBP, Week 20: number analyzed (Participants) | 23 | 8 | 12
  SBP, Week 20 | 1.7 (17.80) | -11.5 (14.69) | -13.8 (25.15)
  SBP, Week 24: number analyzed (Participants) | 21 | 10 | 6
  SBP, Week 24 | 2.9 (13.87) | -1.8 (11.81) | -7.8 (26.06)
  SBP, Week 28: number analyzed (Participants) | 17 | 7 | 5
  SBP, Week 28 | 2.3 (19.10) | -5.7 (20.38) | -5.2 (10.71)
  SBP, Week 32: number analyzed (Participants) | 16 | 8 | 3
  SBP, Week 32 | 3.2 (23.11) | -16.4 (10.03) | -6.3 (5.51)
  SBP, Week 36: number analyzed (Participants) | 13 | 7 | 3
  SBP, Week 36 | 1.6 (15.85) | -8.7 (12.19) | -26.7 (37.75)
  SBP, Week 40: number analyzed (Participants) | 12 | 7 | 2
  SBP, Week 40 | -2.2 (24.44) | -3.4 (9.62) | -34.0 (38.18)
  SBP, Week 44: number analyzed (Participants) | 11 | 6 | 2
  SBP, Week 44 | 2.7 (14.47) | -3.8 (9.83) | -38.0 (32.53)
  SBP, Week 48: number analyzed (Participants) | 11 | 6 | 1
  SBP, Week 48 | 6.5 (18.76) | -6.7 (11.18) | -84.0 (NA) — NA: Data not available as the sample size is 1.
  SBP, Week 52: number analyzed (Participants) | 9 | 5 | 0
  SBP, Week 52 | 7.7 (14.47) | -3.8 (24.78) |
  SBP, Week 56: number analyzed (Participants) | 9 | 5 | 0
  SBP, Week 56 | 8.4 (13.53) | -8.2 (18.74) |
  SBP, Week 60: number analyzed (Participants) | 10 | 4 | 0
  SBP, Week 60 | 9.3 (22.07) | -17.0 (9.31) |
  SBP, Week 64: number analyzed (Participants) | 10 | 4 | 0
  SBP, Week 64 | 3.5 (16.53) | -11.3 (11.24) |
  SBP, Week 68: number analyzed (Participants) | 7 | 2 | 0
  SBP, Week 68 | 0.1 (10.71) | -6.5 (12.02) |
  SBP, Week 72: number analyzed (Participants) | 7 | 1 | 0
  SBP, Week 72 | 7.1 (13.25) | -20.0 (NA) — NA: Data not available as the sample size is 1. |
  SBP, Week 76: number analyzed (Participants) | 6 | 0 | 0
  SBP, Week 76 | 4.5 (12.96) |  |
  SBP, Week 80: number analyzed (Participants) | 6 | 0 | 0
  SBP, Week 80 | 8.7 (6.92) |  |
  SBP, Week 84: number analyzed (Participants) | 6 | 0 | 0
  SBP, Week 84 | 7.0 (20.20) |  |
  SBP, Week 88: number analyzed (Participants) | 6 | 0 | 0
  SBP, Week 88 | -2.7 (16.32) |  |
  SBP, Week 92: number analyzed (Participants) | 5 | 0 | 0
  SBP, Week 92 | 10.4 (16.59) |  |
  SBP, Week 96: number analyzed (Participants) | 4 | 0 | 0
  SBP, Week 96 | -0.5 (4.12) |  |
  SBP, Week 100: number analyzed (Participants) | 5 | 0 | 0
  SBP, Week 100 | 10.8 (7.53) |  |
  SBP, Week 104: number analyzed (Participants) | 5 | 0 | 0
  SBP, Week 104 | 7.0 (16.00) |  |
  SBP, Week 108: number analyzed (Participants) | 5 | 0 | 0
  SBP, Week 108 | 4.6 (7.89) |  |
  SBP, Week 112: number analyzed (Participants) | 4 | 0 | 0
  SBP, Week 112 | 12.3 (10.72) |  |
  SBP, Week 116: number analyzed (Participants) | 4 | 0 | 0
  SBP, Week 116 | 9.3 (15.22) |  |
  SBP, Week 120: number analyzed (Participants) | 3 | 0 | 0
  SBP, Week 120 | 13.3 (19.86) |  |
  SBP, Week 124: number analyzed (Participants) | 3 | 0 | 0
  SBP, Week 124 | 7.3 (8.50) |  |
  SBP, Week 128: number analyzed (Participants) | 2 | 0 | 0
  SBP, Week 128 | -11.0 (9.90) |  |
  SBP, Week 132: number analyzed (Participants) | 2 | 0 | 0
  SBP, Week 132 | -10.5 (10.61) |  |
  SBP, Week 136: number analyzed (Participants) | 2 | 0 | 0
  SBP, Week 136 | -4.0 (18.38) |  |
  SBP, Week 140: number analyzed (Participants) | 2 | 0 | 0
  SBP, Week 140 | 4.5 (23.33) |  |
  SBP, Week 144: number analyzed (Participants) | 1 | 0 | 0
  SBP, Week 144 | 10.0 (0) |  |
  SBP, Week 148: number analyzed (Participants) | 1 | 0 | 0
  SBP, Week 148 | 25.0 (NA) — NA: Data not available as the sample size is 1. |  |
  SBP, Withdrawal/Study Conclusion: number analyzed (Participants) | 23 | 10 | 8
  SBP, Withdrawal/Study Conclusion | 0.5 (16.13) | -1.3 (15.64) | 7.0 (20.28)
  SBP, 30 Day Follow-up: number analyzed (Participants) | 25 | 9 | 5
  SBP, 30 Day Follow-up | 2.4 (19.18) | -3.9 (17.03) | 13.8 (19.25)
  DBP, Week 4: number analyzed (Participants) | 28 | 12 | 18
  DBP, Week 4 | -2.5 (10.36) | -3.9 (10.50) | -4.8 (11.10)
  DBP, Week 8: number analyzed (Participants) | 27 | 13 | 17
  DBP, Week 8 | -0.6 (11.41) | -8.9 (11.54) | -1.2 (12.46)
  DBP, Week 12: number analyzed (Participants) | 24 | 12 | 16
  DBP, Week 12 | -0.3 (10.19) | -6.2 (10.37) | -4.2 (12.87)
  DBP, Week 16: number analyzed (Participants) | 23 | 11 | 15
  DBP, Week 16 | -3.4 (12.98) | -3.2 (8.42) | -4.4 (15.18)
  DBP, Week 20: number analyzed (Participants) | 23 | 8 | 12
  DBP, Week 20 | -3.0 (12.65) | -1.6 (9.53) | -9.1 (13.65)
  DBP, Week 24: number analyzed (Participants) | 21 | 10 | 6
  DBP, Week 24 | -1.2 (11.30) | -1.8 (6.56) | -5.2 (13.08)
  DBP, Week 28: number analyzed (Participants) | 17 | 7 | 5
  DBP, Week 28 | -1.8 (14.27) | -2.1 (8.15) | -2.0 (5.05)
  DBP, Week 32: number analyzed (Participants) | 16 | 8 | 3
  DBP, Week 32 | -2.2 (13.70) | -6.3 (10.24) | -4.7 (6.51)
  DBP, Week 36: number analyzed (Participants) | 13 | 7 | 3
  DBP, Week 36 | -7.2 (6.48) | -3.3 (6.40) | -10.7 (11.02)
  DBP, Week 40: number analyzed (Participants) | 12 | 7 | 2
  DBP, Week 40 | -9.3 (11.36) | -0.7 (13.76) | -8.0 (19.80)
  DBP, Week 44: number analyzed (Participants) | 11 | 6 | 2
  DBP, Week 44 | -9.0 (6.59) | -2.3 (10.33) | -19.5 (6.36)
  DBP, Week 48: number analyzed (Participants) | 11 | 6 | 1
  DBP, Week 48 | -3.9 (7.57) | -0.2 (8.13) | -34.0 (NA) — NA: Data not available as the sample size is 1
  DBP, Week 52: number analyzed (Participants) | 9 | 5 | 0
  DBP, Week 52 | -7.4 (13.46) | -3.0 (12.33) |
  DBP, Week 56: number analyzed (Participants) | 9 | 5 | 0
  DBP, Week 56 | -5.1 (8.62) | -3.4 (7.99) |
  DBP, Week 60: number analyzed (Participants) | 10 | 4 | 0
  DBP, Week 60 | -3.6 (11.56) | -6.3 (6.24) |
  DBP, Week 64: number analyzed (Participants) | 10 | 4 | 0
  DBP, Week 64 | -7.7 (12.27) | -5.3 (8.54) |
  DBP, Week 68: number analyzed (Participants) | 7 | 2 | 0
  DBP, Week 68 | -11.0 (6.40) | -3.5 (7.78) |
  DBP, Week 72: number analyzed (Participants) | 7 | 1 | 0
  DBP, Week 72 | 3.0 (9.26) | -16.0 (NA) — NA: Data not available as the sample size is 1. |
  DBP, Week 76: number analyzed (Participants) | 6 | 0 | 0
  DBP, Week 76 | -4.8 (5.00) |  |
  DBP, Week 80: number analyzed (Participants) | 6 | 0 | 0
  DBP, Week 80 | -3.5 (5.58) |  |
  DBP, Week 84: number analyzed (Participants) | 6 | 0 | 0
  DBP, Week 84 | -5.8 (9.50) |  |
  DBP, Week 88: number analyzed (Participants) | 6 | 0 | 0
  DBP, Week 88 | -9.3 (11.48) |  |
  DBP, Week 92: number analyzed (Participants) | 5 | 0 | 0
  DBP, Week 92 | -3.8 (5.26) |  |
  DBP, Week 96: number analyzed (Participants) | 4 | 0 | 0
  DBP, Week 96 | -7.3 (6.29) |  |
  DBP, Week 100: number analyzed (Participants) | 5 | 0 | 0
  DBP, Week 100 | -4.4 (6.50) |  |
  DBP, Week 104: number analyzed (Participants) | 5 | 0 | 0
  DBP, Week 104 | -4.6 (9.10) |  |
  DBP, Week 108: number analyzed (Participants) | 5 | 0 | 0
  DBP, Week 108 | -2.0 (5.89) |  |
  DBP, Week 116: number analyzed (Participants) | 4 | 0 | 0
  DBP, Week 116 | -8.5 (9.33) |  |
  DBP, Week 120: number analyzed (Participants) | 3 | 0 | 0
  DBP, Week 120 | -6.0 (7.94) |  |
  DBP, Week 124: number analyzed (Participants) | 3 | 0 | 0
  DBP, Week 124 | -6.0 (6.00) |  |
  DBP, Week 128: number analyzed (Participants) | 2 | 0 | 0
  DBP, Week 128 | -12.5 (0.71) |  |
  DBP, Week 132: number analyzed (Participants) | 2 | 0 | 0
  DBP, Week 132 | -14.5 (4.95) |  |
  DBP, Week 136: number analyzed (Participants) | 2 | 0 | 0
  DBP, Week 136 | -17.0 (4.24) |  |
  DBP, Week 140: number analyzed (Participants) | 2 | 0 | 0
  DBP, Week 140 | -7.5 (10.61) |  |
  DBP, Week 144: number analyzed (Participants) | 1 | 0 | 0
  DBP, Week 144 | 0.0 (0) |  |
  DBP, Week 148: number analyzed (Participants) | 1 | 0 | 0
  DBP, Week 148 | 1.0 (NA) — NA: Data not available as the sample size is 1. |  |
  DBP, Withdrawal/Study Conclusion: number analyzed (Participants) | 23 | 10 | 8
  DBP, Withdrawal/Study Conclusion | -0.5 (11.39) | -0.4 (12.08) | 2.1 (8.64)
  DBP, 30 Day Follow-up: number analyzed (Participants) | 25 | 9 | 5
  DBP, 30 Day Follow-up | -0.8 (11.96) | 0.8 (11.62) | 3.2 (9.98)

11. Primary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Heart rate was measured at Baseline and every 4 weeks thereafter up to withdrawal/study completion and at the 30 day follow-up visit. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population. Safety Population: all participants who were randomized and received at least one dose of investigational product.
  Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Beats per minute (BPM)
  Week 4: number analyzed (Participants) | 28 | 12 | 18
  Week 4 | -1.714 (10.9099) | -3.417 (26.3593) | 3.333 (12.1268)
  Week 8: number analyzed (Participants) | 27 | 13 | 17
  Week 8 | -5.667 (14.7908) | -3.231 (16.8481) | 5.353 (10.7642)
  Week 12: number analyzed (Participants) | 23 | 12 | 16
  Week 12 | -0.217 (10.7109) | -0.417 (15.6812) | -2.875 (10.6074)
  Week 16: number analyzed (Participants) | 22 | 11 | 14
  Week 16 | -0.478 (13.4667) | 2.625 (15.1369) | -1.917 (10.9084)
  Week 24: number analyzed (Participants) | 21 | 10 | 6
  Week 24 | -0.476 (16.7768) | -5.300 (15.1808) | 5.167 (10.2843)
  Week 28: number analyzed (Participants) | 16 | 7 | 5
  Week 28 | -4.313 (16.0155) | -1.429 (17.7281) | 3.600 (8.5615)
  Week 32: number analyzed (Participants) | 15 | 8 | 3
  Week 32 | -4.933 (16.6496) | -0.500 (11.1098) | 0.333 (10.5987)
  Week 36: number analyzed (Participants) | 13 | 7 | 3
  Week 36 | -5.000 (13.0128) | 4.857 (18.4791) | 7.000 (11.5326)
  Week 40: number analyzed (Participants) | 12 | 7 | 2
  Week 40 | -1.000 (14.1614) | -3.571 (17.6149) | -2.500 (9.1924)
  Week 44: number analyzed (Participants) | 11 | 6 | 2
  Week 44 | -3.000 (11.1624) | -5.000 (17.9778) | -0.500 (10.6066)
  Week 48: number analyzed (Participants) | 10 | 6 | 1
  Week 48 | -5.500 (8.1955) | -2.500 (12.9422) | -14.000 (NA) — NA: Data not available as the sample size is 1
  Week 52: number analyzed (Participants) | 9 | 5 | 0
  Week 52 | -1.889 (14.4866) | -2.000 (11.8533) |
  Week 56: number analyzed (Participants) | 8 | 5 | 0
  Week 56 | -2.000 (13.4907) | -2.000 (15.2151) |
  Week 60: number analyzed (Participants) | 10 | 4 | 0
  Week 60 | -2.600 (13.3766) | 1.500 (15.0222) |
  Week 64: number analyzed (Participants) | 9 | 4 | 0
  Week 64 | -4.667 (16.1245) | 0.000 (15.3840) |
  Week 68: number analyzed (Participants) | 7 | 2 | 0
  Week 68 | -8.286 (21.1638) | 1.000 (25.4558) |
  Week 72: number analyzed (Participants) | 7 | 1 | 0
  Week 72 | -0.714 (21.0295) | 19.000 (NA) — NA: Data not available as the sample size is 1. |
  Week 76: number analyzed (Participants) | 6 | 0 | 0
  Week 76 | -0.500 (16.6463) |  |
  Week 80: number analyzed (Participants) | 5 | 0 | 0
  Week 80 | 0.800 (14.4810) |  |
  Week 84: number analyzed (Participants) | 5 | 0 | 0
  Week 84 | 9.200 (21.1234) |  |
  Week 88: number analyzed (Participants) | 5 | 0 | 0
  Week 88 | 2.200 (24.6110) |  |
  Week 92: number analyzed (Participants) | 5 | 0 | 0
  Week 92 | -2.400 (10.1390) |  |
  Week 96: number analyzed (Participants) | 4 | 0 | 0
  Week 96 | -8.250 (7.6322) |  |
  Week 100: number analyzed (Participants) | 4 | 0 | 0
  Week 100 | -6.750 (13.1751) |  |
  Week 104: number analyzed (Participants) | 5 | 0 | 0
  Week 104 | -6.800 (15.3525) |  |
  Week 108: number analyzed (Participants) | 4 | 0 | 0
  Week 108 | -8.750 (6.4485) |  |
  Week 112: number analyzed (Participants) | 3 | 0 | 0
  Week 112 | -0.667 (15.0444) |  |
  Week 116: number analyzed (Participants) | 3 | 0 | 0
  Week 116 | -4.667 (14.5717) |  |
  Week 120: number analyzed (Participants) | 3 | 0 | 0
  Week 120 | -7.667 (9.4516) |  |
  Week 124: number analyzed (Participants) | 3 | 0 | 0
  Week 124 | -5.333 (13.2035) |  |
  Week 128: number analyzed (Participants) | 2 | 0 | 0
  Week 128 | 1.000 (21.2132) |  |
  Week 132: number analyzed (Participants) | 2 | 0 | 0
  Week 132 | -4.000 (14.1421) |  |
  Week 136: number analyzed (Participants) | 2 | 0 | 0
  Week 136 | -4.000 (15.5563) |  |
  Week 140: number analyzed (Participants) | 2 | 0 | 0
  Week 140 | -3.500 (16.2635) |  |
  Week 144: number analyzed (Participants) | 1 | 0 | 0
  Week 144 | 3.000 (NA) — NA: Data not available as the sample size is 1. |  |
  Week 148: number analyzed (Participants) | 1 | 0 | 0
  Week 148 | 6.000 (NA) — NA: Data not available as the sample size is 1. |  |
  Withdrawal/Study Conclusion: number analyzed (Participants) | 23 | 10 | 8
  Withdrawal/Study Conclusion | -1.435 (19.3481) | -7.900 (19.3990) | 7.750 (9.8814)
  30 Day Follow-up: number analyzed (Participants) | 25 | 9 | 5
  30 Day Follow-up | 0.560 (13.1564) | -7.889 (17.3526) | 13.200 (11.6060)

12. Primary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points
Description: Body temperature was measured at Baseline and every 4 weeks thereafter up to withdrawal/study completion and at the 30 day follow-up visit. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Degree Celsius
  Week 4: number analyzed (Participants) | 28 | 12 | 18
  Week 4 | -0.229 (0.5062) | -0.242 (0.3605) | 0.078 (0.5976)
  Week 8: number analyzed (Participants) | 27 | 13 | 17
  Week 8 | 0.011 (0.5250) | -0.154 (0.4294) | 0.247 (0.4652)
  Week 12: number analyzed (Participants) | 24 | 12 | 15
  Week 12 | 0.021 (0.4374) | -0.567 (0.4960) | 0.173 (0.4636)
  Week 16: number analyzed (Participants) | 23 | 11 | 14
  Week 16 | -0.052 (0.5814) | -0.127 (0.4880) | 0.121 (0.5494)
  Week 20: number analyzed (Participants) | 22 | 8 | 12
  Week 20 | 0.018 (0.5712) | -0.238 (0.4138) | 0.300 (0.3536)
  Week 24: number analyzed (Participants) | 21 | 9 | 6
  Week 24 | 0.157 (0.5006) | -0.100 (0.4138) | 0.017 (0.5193)
  Week 28: number analyzed (Participants) | 17 | 7 | 5
  Week 28 | -0.094 (0.4956) | -0.529 (0.4751) | 0.300 (0.3536)
  Week 32: number analyzed (Participants) | 16 | 8 | 3
  Week 32 | -0.156 (0.6077) | -0.237 (0.2134) | 0.000 (0.2000)
  Week 36: number analyzed (Participants) | 13 | 7 | 3
  Week 36 | -0.215 (0.5728) | -0.129 (0.3946) | 0.533 (0.3786)
  Week 40: number analyzed (Participants) | 11 | 7 | 2
  Week 40 | 0.045 (0.4634) | -0.314 (0.1952) | 0.450 (0.9192)
  Week 44: number analyzed (Participants) | 11 | 6 | 2
  Week 44 | -0.182 (0.4729) | -0.217 (0.3920) | 0.250 (0.0707)
  Week 48: number analyzed (Participants) | 11 | 6 | 1
  Week 48 | -0.109 (0.4571) | -0.200 (0.1414) | 0.300 (NA) — NA: Data not available as the sample size is 1.
  Week 52: number analyzed (Participants) | 9 | 5 | 0
  Week 52 | -0.222 (1.0616) | -0.340 (0.3286) |
  Week 56: number analyzed (Participants) | 9 | 5 | 0
  Week 56 | 0.111 (0.6489) | -0.240 (0.6427) |
  Week 60: number analyzed (Participants) | 10 | 4 | 0
  Week 60 | -0.070 (0.5889) | -0.225 (0.2754) |
  Week 64: number analyzed (Participants) | 10 | 4 | 0
  Week 64 | -0.080 (0.4662) | -0.150 (0.1732) |
  Week 68: number analyzed (Participants) | 7 | 2 | 0
  Week 68 | 0.286 (0.6744) | -0.550 (0.0707) |
  Week 72: number analyzed (Participants) | 7 | 1 | 0
  Week 72 | 0.057 (0.7390) | -0.400 (NA) — NA: Data not available as the sample size is 1. |
  Week 76: number analyzed (Participants) | 6 | 0 | 0
  Week 76 | 0.017 (0.4834) |  |
  Week 80: number analyzed (Participants) | 6 | 0 | 0
  Week 80 | -0.150 (0.6442) |  |
  Week 84: number analyzed (Participants) | 6 | 0 | 0
  Week 84 | 0.067 (0.5610) |  |
  Week 88: number analyzed (Participants) | 6 | 0 | 0
  Week 88 | -0.267 (0.4131) |  |
  Week 92: number analyzed (Participants) | 5 | 0 | 0
  Week 92 | -0.200 (0.8155) |  |
  Week 96: number analyzed (Participants) | 4 | 0 | 0
  Week 96 | -0.125 (0.4573) |  |
  Week 100: number analyzed (Participants) | 5 | 0 | 0
  Week 100 | -0.100 (0.9083) |  |
  Week 104: number analyzed (Participants) | 5 | 0 | 0
  Week 104 | -0.160 (0.7436) |  |
  Week 108: number analyzed (Participants) | 4 | 0 | 0
  Week 108 | 0.080 (0.6099) |  |
  Week 112: number analyzed (Participants) | 4 | 0 | 0
  Week 112 | 0.050 (0.5000) |  |
  Week 116: number analyzed (Participants) | 3 | 0 | 0
  Week 116 | 0.250 (0.6403) |  |
  Week 120: number analyzed (Participants) | 3 | 0 | 0
  Week 120 | 0.200 (0.4359) |  |
  Week 124: number analyzed (Participants) | 3 | 0 | 0
  Week 124 | 0.167 (0.8083) |  |
  Week 128: number analyzed (Participants) | 2 | 0 | 0
  Week 128 | 0.200 (1.4142) |  |
  Week 132: number analyzed (Participants) | 2 | 0 | 0
  Week 132 | -0.150 (1.2021) |  |
  Week 136: number analyzed (Participants) | 2 | 0 | 0
  Week 136 | 0.000 (1.2728) |  |
  Week 140: number analyzed (Participants) | 2 | 0 | 0
  Week 140 | 0.450 (1.3435) |  |
  Week 144: number analyzed (Participants) | 1 | 0 | 0
  Week 144 | 1.300 (NA) — NA: Data not available as the sample size is 1. |  |
  Week 148: number analyzed (Participants) | 1 | 0 | 0
  Week 148 | 0.700 (NA) — NA: Data not available as the sample size is 1. |  |
  Withdrawal/Study Conclusion: number analyzed (Participants) | 23 | 10 | 8
  Withdrawal/Study Conclusion | -0.083 (0.6833) | -0.020 (0.4367) | 0.237 (0.5999)
  30 Day Follow-up: number analyzed (Participants) | 25 | 9 | 5
  30 Day Follow-up | -0.092 (0.6238) | -0.400 (0.5074) | 0.140 (0.5320)

13. Primary Outcome: Number of Participants With at Least 1 Event of Left Ventricular Ejection Fraction Decrease With the Indicated Characteristics
Description: Events of left ventricular ejection fraction (LVEF) decrease were based on the number of participants who had an actual event and was characterized as serious, related to investigational product, leading to withdrawal from the study and/or fatal.
Time Frame: Baseline and every 8 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population. Only the participants with at least one of event of LVEF decrease were analyzed.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants | 8 | 2 | 0

14. Primary Outcome: Number of Participants With the Indicated Eastern Cooperative Oncology Group (ECOG) Performance Status Value
Description: The Eastern Cooperative Oncology Group (ECOG) performance status scales and grades/criteria are used to assess how a participant's disease is progressing, to assess how the disease affects the daily living abilities of the participant, and to determine appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. Grade 5, dead.
Time Frame: Baseline and every 4 weeks thereafter up to withdrawal/study completion and 30 day follow-up, up to approx. 3.5 years
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the safety population.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants
  Screening, Grade 3 | 0 | 0 | 0
  Screening, Grade 4 | 0 | 0 | 0
  Screening, Grade 5 | 0 | 0 | 0
  Day 1 pre-dose, Grade 3: number analyzed (Participants) | 29 | 13 | 20
  Day 1 pre-dose, Grade 3 | 0 | 0 | 0
  Day 1 pre-dose, Grade 4: number analyzed (Participants) | 29 | 13 | 20
  Day 1 pre-dose, Grade 4 | 0 | 0 | 0
  Day 1 pre-dose, Grade 5: number analyzed (Participants) | 29 | 13 | 20
  Day 1 pre-dose, Grade 5 | 0 | 0 | 0
  Week 4, Grade 3: number analyzed (Participants) | 28 | 12 | 18
  Week 4, Grade 3 | 0 | 0 | 0
  Week 4, Grade 4: number analyzed (Participants) | 28 | 12 | 18
  Week 4, Grade 4 | 0 | 0 | 0
  Week 4, Grade 5: number analyzed (Participants) | 28 | 12 | 18
  Week 4, Grade 5 | 0 | 0 | 0
  Week 8, Grade 3: number analyzed (Participants) | 27 | 13 | 16
  Week 8, Grade 3 | 0 | 0 | 0
  Week 8, Grade 4: number analyzed (Participants) | 27 | 13 | 16
  Week 8, Grade 4 | 0 | 0 | 0
  Week 8, Grade 5: number analyzed (Participants) | 27 | 13 | 16
  Week 8, Grade 5 | 0 | 0 | 0
  Week 12, Grade 3: number analyzed (Participants) | 24 | 12 | 16
  Week 12, Grade 3 | 0 | 0 | 0
  Week 12, Grade 4: number analyzed (Participants) | 24 | 12 | 16
  Week 12, Grade 4 | 0 | 0 | 0
  Week 12, Grade 5: number analyzed (Participants) | 24 | 12 | 16
  Week 12, Grade 5 | 0 | 0 | 0
  Week 16, Grade 3: number analyzed (Participants) | 22 | 11 | 15
  Week 16, Grade 3 | 0 | 0 | 0
  Week 16, Grade 4: number analyzed (Participants) | 22 | 11 | 15
  Week 16, Grade 4 | 0 | 0 | 0
  Week 16, Grade 5: number analyzed (Participants) | 22 | 11 | 15
  Week 16, Grade 5 | 0 | 0 | 0
  Week 20, Grade 3: number analyzed (Participants) | 24 | 10 | 11
  Week 20, Grade 3 | 0 | 0 | 0
  Week 20, Grade 4: number analyzed (Participants) | 24 | 10 | 11
  Week 20, Grade 4 | 0 | 0 | 0
  Week 20, Grade 5: number analyzed (Participants) | 24 | 10 | 11
  Week 20, Grade 5 | 0 | 0 | 0
  Week 24, Grade 3: number analyzed (Participants) | 21 | 10 | 6
  Week 24, Grade 3 | 0 | 0 | 0
  Week 24, Grade 4: number analyzed (Participants) | 21 | 10 | 6
  Week 24, Grade 4 | 0 | 0 | 0
  Week 24, Grade 5: number analyzed (Participants) | 21 | 10 | 6
  Week 24, Grade 5 | 0 | 0 | 0
  Week 28, Grade 3: number analyzed (Participants) | 17 | 8 | 4
  Week 28, Grade 3 | 0 | 0 | 0
  Week 28, Grade 4: number analyzed (Participants) | 17 | 8 | 4
  Week 28, Grade 4 | 0 | 0 | 0
  Week 28, Grade 5: number analyzed (Participants) | 17 | 8 | 4
  Week 28, Grade 5 | 0 | 0 | 0
  Week 32, Grade 3: number analyzed (Participants) | 16 | 8 | 3
  Week 32, Grade 3 | 0 | 0 | 0
  Week 32, Grade 4: number analyzed (Participants) | 16 | 8 | 3
  Week 32, Grade 4 | 0 | 0 | 0
  Week 32, Grade 5: number analyzed (Participants) | 16 | 8 | 3
  Week 32, Grade 5 | 0 | 0 | 0
  Week 36, Grade 3: number analyzed (Participants) | 12 | 7 | 3
  Week 36, Grade 3 | 0 | 0 | 0
  Week 36, Grade 4: number analyzed (Participants) | 12 | 7 | 3
  Week 36, Grade 4 | 0 | 0 | 0
  Week 36, Grade 5: number analyzed (Participants) | 12 | 7 | 3
  Week 36, Grade 5 | 0 | 0 | 0
  Week 40, Grade 3: number analyzed (Participants) | 12 | 7 | 2
  Week 40, Grade 3 | 0 | 0 | 0
  Week 40, Grade 4: number analyzed (Participants) | 12 | 7 | 2
  Week 40, Grade 4 | 0 | 0 | 0
  Week 40, Grade 5: number analyzed (Participants) | 12 | 7 | 2
  Week 40, Grade 5 | 0 | 0 | 0
  Week 44, Grade 3: number analyzed (Participants) | 11 | 6 | 2
  Week 44, Grade 3 | 0 | 0 | 0
  Week 44, Grade 4: number analyzed (Participants) | 11 | 6 | 2
  Week 44, Grade 4 | 0 | 0 | 0
  Week 44, Grade 5: number analyzed (Participants) | 11 | 6 | 2
  Week 44, Grade 5 | 0 | 0 | 0
  Week 48, Grade 3: number analyzed (Participants) | 10 | 6 | 1
  Week 48, Grade 3 | 0 | 0 | 0
  Week 48, Grade 4: number analyzed (Participants) | 10 | 6 | 1
  Week 48, Grade 4 | 0 | 0 | 0
  Week 48, Grade 5: number analyzed (Participants) | 10 | 6 | 1
  Week 48, Grade 5 | 0 | 0 | 0
  Week 52, Grade3: number analyzed (Participants) | 9 | 5 | 0
  Week 52, Grade3 | 0 | 0 |
  Week 52, Grade4: number analyzed (Participants) | 9 | 5 | 0
  Week 52, Grade4 | 0 | 0 |
  Week 52, Grade5: number analyzed (Participants) | 9 | 5 | 0
  Week 52, Grade5 | 0 | 0 |
  Week 56, Grade 3: number analyzed (Participants) | 8 | 4 | 0
  Week 56, Grade 3 | 0 | 0 |
  Week 56, Grade 4: number analyzed (Participants) | 8 | 4 | 0
  Week 56, Grade 4 | 0 | 0 |
  Week 56, Grade 5: number analyzed (Participants) | 8 | 4 | 0
  Week 56, Grade 5 | 0 | 0 |
  Week 60, Grade 3: number analyzed (Participants) | 10 | 4 | 0
  Week 60, Grade 3 | 0 | 0 |
  Week 60, Grade 4: number analyzed (Participants) | 10 | 4 | 0
  Week 60, Grade 4 | 0 | 0 |
  Week 60, Grade 5: number analyzed (Participants) | 10 | 4 | 0
  Week 60, Grade 5 | 0 | 0 |
  Week 64, Grade 3: number analyzed (Participants) | 9 | 4 | 0
  Week 64, Grade 3 | 0 | 0 |
  Week 64, Grade 4: number analyzed (Participants) | 9 | 4 | 0
  Week 64, Grade 4 | 0 | 0 |
  Week 64, Grade 5: number analyzed (Participants) | 9 | 4 | 0
  Week 64, Grade 5 | 0 | 0 |
  Week 68, Grade3: number analyzed (Participants) | 8 | 2 | 0
  Week 68, Grade3 | 0 | 0 |
  Week 68, Grade4: number analyzed (Participants) | 8 | 2 | 0
  Week 68, Grade4 | 0 | 0 |
  Week 68, Grade5: number analyzed (Participants) | 8 | 2 | 0
  Week 68, Grade5 | 0 | 0 |
  Week 72, Grade 3: number analyzed (Participants) | 7 | 1 | 0
  Week 72, Grade 3 | 0 | 0 |
  Week 72, Grade 4: number analyzed (Participants) | 7 | 1 | 0
  Week 72, Grade 4 | 0 | 0 |
  Week 72, Grade 5: number analyzed (Participants) | 7 | 1 | 0
  Week 72, Grade 5 | 0 | 0 |
  Week 76, Grade3: number analyzed (Participants) | 6 | 0 | 0
  Week 76, Grade3 | 0 |  |
  Week 76, Grade4: number analyzed (Participants) | 6 | 0 | 0
  Week 76, Grade4 | 0 |  |
  Week 76, Grade5: number analyzed (Participants) | 6 | 0 | 0
  Week 76, Grade5 | 0 |  |
  Week 80, Grade 3: number analyzed (Participants) | 6 | 0 | 0
  Week 80, Grade 3 | 0 |  |
  Week 80, Grade 4: number analyzed (Participants) | 6 | 0 | 0
  Week 80, Grade 4 | 0 |  |
  Week 80, Grade 5: number analyzed (Participants) | 6 | 0 | 0
  Week 80, Grade 5 | 0 |  |
  Week 84, Grade 3: number analyzed (Participants) | 6 | 0 | 0
  Week 84, Grade 3 | 0 |  |
  Week 84, Grade 4: number analyzed (Participants) | 6 | 0 | 0
  Week 84, Grade 4 | 0 |  |
  Week 84, Grade 5: number analyzed (Participants) | 6 | 0 | 0
  Week 84, Grade 5 | 0 |  |
  Week 88, Grade 3: number analyzed (Participants) | 6 | 0 | 0
  Week 88, Grade 3 | 0 |  |
  Week 88, Grade 4: number analyzed (Participants) | 6 | 0 | 0
  Week 88, Grade 4 | 0 |  |
  Week 88, Grade 5: number analyzed (Participants) | 6 | 0 | 0
  Week 88, Grade 5 | 0 |  |
  Week 92, Grade 3: number analyzed (Participants) | 5 | 0 | 0
  Week 92, Grade 3 | 0 |  |
  Week 92, Grade 4: number analyzed (Participants) | 5 | 0 | 0
  Week 92, Grade 4 | 0 |  |
  Week 92, Grade 5: number analyzed (Participants) | 5 | 0 | 0
  Week 92, Grade 5 | 0 |  |
  Week 96, Grade 3: number analyzed (Participants) | 4 | 0 | 0
  Week 96, Grade 3 | 0 |  |
  Week 96, Grade 4: number analyzed (Participants) | 4 | 0 | 0
  Week 96, Grade 4 | 0 |  |
  Week 96, Grade 5: number analyzed (Participants) | 4 | 0 | 0
  Week 96, Grade 5 | 0 |  |
  Week 100, Grade 3: number analyzed (Participants) | 5 | 0 | 0
  Week 100, Grade 3 | 0 |  |
  Week 100, Grade 4: number analyzed (Participants) | 5 | 0 | 0
  Week 100, Grade 4 | 0 |  |
  Week 100, Grade 5: number analyzed (Participants) | 5 | 0 | 0
  Week 100, Grade 5 | 0 |  |
  Week 104, Grade 3: number analyzed (Participants) | 5 | 0 | 0
  Week 104, Grade 3 | 0 |  |
  Week 104, Grade 4: number analyzed (Participants) | 5 | 0 | 0
  Week 104, Grade 4 | 0 |  |
  Week 104, Grade 5: number analyzed (Participants) | 5 | 0 | 0
  Week 104, Grade 5 | 0 |  |
  Week 108, Grade 3: number analyzed (Participants) | 5 | 0 | 0
  Week 108, Grade 3 | 0 |  |
  Week 108, Grade 4: number analyzed (Participants) | 5 | 0 | 0
  Week 108, Grade 4 | 0 |  |
  Week 108, Grade 5: number analyzed (Participants) | 5 | 0 | 0
  Week 108, Grade 5 | 0 |  |
  Week 112, Grade 3: number analyzed (Participants) | 4 | 0 | 0
  Week 112, Grade 3 | 0 |  |
  Week 112, Grade 4: number analyzed (Participants) | 4 | 0 | 0
  Week 112, Grade 4 | 0 |  |
  Week 112, Grade 5: number analyzed (Participants) | 4 | 0 | 0
  Week 112, Grade 5 | 0 |  |
  Week 116, Grade 3: number analyzed (Participants) | 4 | 0 | 0
  Week 116, Grade 3 | 0 |  |
  Week 116, Grade 4: number analyzed (Participants) | 4 | 0 | 0
  Week 116, Grade 4 | 0 |  |
  Week 116, Grade 5: number analyzed (Participants) | 4 | 0 | 0
  Week 116, Grade 5 | 0 |  |
  Week 120, Grade 3: number analyzed (Participants) | 3 | 0 | 0
  Week 120, Grade 3 | 0 |  |
  Week 120, Grade 4: number analyzed (Participants) | 3 | 0 | 0
  Week 120, Grade 4 | 0 |  |
  Week 120, Grade 5: number analyzed (Participants) | 3 | 0 | 0
  Week 120, Grade 5 | 0 |  |
  Week 124, Grade 3: number analyzed (Participants) | 3 | 0 | 0
  Week 124, Grade 3 | 0 |  |
  Week 124, Grade 4: number analyzed (Participants) | 3 | 0 | 0
  Week 124, Grade 4 | 0 |  |
  Week 124, Grade 5: number analyzed (Participants) | 3 | 0 | 0
  Week 124, Grade 5 | 0 |  |
  Week 128, Grade 3: number analyzed (Participants) | 2 | 0 | 0
  Week 128, Grade 3 | 0 |  |
  Week 128, Grade 4: number analyzed (Participants) | 2 | 0 | 0
  Week 128, Grade 4 | 0 |  |
  Week 128, Grade 5: number analyzed (Participants) | 2 | 0 | 0
  Week 128, Grade 5 | 0 |  |
  Week 132, Grade 3: number analyzed (Participants) | 2 | 0 | 0
  Week 132, Grade 3 | 0 |  |
  Week 132, Grade 4: number analyzed (Participants) | 2 | 0 | 0
  Week 132, Grade 4 | 0 |  |
  Week 132, Grade 5: number analyzed (Participants) | 2 | 0 | 0
  Week 132, Grade 5 | 0 |  |
  Week 136, Grade 3: number analyzed (Participants) | 2 | 0 | 0
  Week 136, Grade 3 | 0 |  |
  Week 136, Grade 4: number analyzed (Participants) | 2 | 0 | 0
  Week 136, Grade 4 | 0 |  |
  Week 136, Grade 5: number analyzed (Participants) | 2 | 0 | 0
  Week 136, Grade 5 | 0 |  |
  Week 140, Grade 3: number analyzed (Participants) | 2 | 0 | 0
  Week 140, Grade 3 | 2 |  |
  Week 140, Grade 4: number analyzed (Participants) | 2 | 0 | 0
  Week 140, Grade 4 | 0 |  |
  Week 140, Grade 5: number analyzed (Participants) | 2 | 0 | 0
  Week 140, Grade 5 | 0 |  |
  Week 144, Grade 3: number analyzed (Participants) | 1 | 0 | 0
  Week 144, Grade 3 | 0 |  |
  Week 144, Grade 4: number analyzed (Participants) | 1 | 0 | 0
  Week 144, Grade 4 | 0 |  |
  Week 144, Grade 5: number analyzed (Participants) | 1 | 0 | 0
  Week 144, Grade 5 | 0 |  |
  Week 148, Grade 3: number analyzed (Participants) | 1 | 0 | 0
  Week 148, Grade 3 | 0 |  |
  Week 148, Grade 4: number analyzed (Participants) | 1 | 0 | 0
  Week 148, Grade 4 | 0 |  |
  Week 148, Grade 5: number analyzed (Participants) | 1 | 0 | 0
  Week 148, Grade 5 | 0 |  |
  Withdrawal/Study conclusion, Grade 3: number analyzed (Participants) | 22 | 10 | 7
  Withdrawal/Study conclusion, Grade 3 | 0 | 0 | 0
  Withdrawal/Study conclusion, Grade 4: number analyzed (Participants) | 22 | 10 | 7
  Withdrawal/Study conclusion, Grade 4 | 0 | 0 | 0
  Withdrawal/Study conclusion, Grade 5: number analyzed (Participants) | 22 | 10 | 7
  Withdrawal/Study conclusion, Grade 5 | 0 | 0 | 0

15. Primary Outcome: Number of Participants Who Received Any Concomitant Medications During the Study Period
Description: Number of participants who received any concomitant medication along with study drugs (lapatinib, trastuzumab and paclitaxel) were counted during the treatment period.
Time Frame: withdrawal/study completion, up to approx. 3.5 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Participants | 29 | 14 | 20

16. Primary Outcome: Overall Response (OR): Percentage of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Confirmed Partial Response (PR) as Assessed by the Investigator
Description: OR is defined as the number of participants achieving either a CR or PR, per Response Evaluation Criteria in Solid Tumors (RECIST). The best OR is defined as the best response recorded from the start of treatment until progressive disease (PD)/recurrence. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s), as assessed by the IRC. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at subsequent assessments made >=28 days after the original response. Participants with an unknown or missing response are treated as non-responders.
Time Frame: From the date of the first dose of investigational product to end of study, up to approx. 7 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Percentage of participants | 79.3 [64.6 to 94.1] | 71.4 [47.8 to 95.1] | 70.0 [49.9 to 90.1]

17. Secondary Outcome: Time to Response as Assessed by the Investigator
Description: Time to Response was defined for subjects who had a confirmed CR or PR as the time from first dose until first documented evidence of partial or complete tumour response (whichever status was recorded first). CR is defined as the disappearance of all TLs & non-TLs. PR is defined as at least a 30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s). PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs.
Time Frame: From the date of the first dose of investigational product until the first documented evidence of a PR or CR, up to approx. 7 years
Population: Safety Population. Safety Population: all participants who were randomized and received at least one dose of investigational product. Only those participants with CR or PR were analyzed.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 23 | 10 | 14
Participants
  Week 8 | 15 | 8 | 8
  Week 12 | 5 | 1 | 1
  Week 16 | 2 | 1 | 3
  Week 20 | 0 | 0 | 1
  Week 24 | 1 | 0 | 0
  Week 28 | 0 | 0 | 1

18. Secondary Outcome: Duration of Response (DoR), as Assessed by the Investigator
Description: DoR is defined for the subset of participants who had a confirmed CR (disappearance of all TLs and non-TLs) or PR (>=30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL[s]) as the time from the first documented evidence of a CR or PR until the first documentation of radiological PD or death due to breast cancer, if sooner. PD is defined as >=20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. For participants who did not progress or die, DoR was censored on the date of the last radiological scan. If a participant had only a Baseline visit or did not have a date of a radiological scan that was later than the date of initiation of anti-cancer therapy, DoR was censored at the start date of treatment.
Time Frame: From the first documented evidence of a PR or CR until the earlier of the date of disease progression or the date of death due to breast cancer, up to approx. 7 years
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Weeks | 56.6 [27.6 to 117.7] | 59.0 [33.1 to 88.7] | 70.6 [31.4 to 103.1]

19. Secondary Outcome: Percentage of Participants With Clinical Benefit (Complete Response (CR), Partial Response (PR), and Stable Disease [SD] for at Least 24 Weeks) as Assessed by Investigator
Description: Clinical benefit is defined as the percentage of participants achieving either a CR or PR or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of the LD of target lesions, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions), taking as reference, the smallest sum LD since the treatment started) for at least 24 weeks. This was based on confirmed responses from the investigator assessment of clinical benefit.
Time Frame: From the date of the first dose of investigational product until the first documented evidence of a PR or CR or SD until the earlier of the date of disease progression or the date of death due to breast cancer, up to approx. 7 years
Population: Safety Population. Safety Population: all participants who were randomized and received at least one dose of investigational product. Only those participants with CR, PR and SD for at least 24 weeks were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Percentage of Participants | 79.3 [64.6 to 94.1] | 71.4 [47.8 to 95.1] | 70.0 [49.9 to 90.1]

20. Secondary Outcome: Progression-free Survival as Assessed by the Investigator
Description: Progression-free survival is defined as the time from randomization until the earliest date of disease progression or death due to any cause, if sooner. Disease progression was based on the investigator's assessments of the objective evidence (e.g., radiological scans and medical photographs). For participants who do not progress, or die, progression-free survival was censored at the time of the last investigator assessed radiological scan preceding the initiation of any alternative anti-cancer therapy. Progression-free survival was summarized using Kaplan-Meier curves.
Time Frame: From the date of the first dose of investigational product until the earlier of the date of disease progression or death due to any cause, up to approx. 7 years
Population: Safety Population: all participants who were randomized and received at least one dose of investigational product. Only those participants with CR, PR and SD for at least 24 weeks were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
Number analyzed (Participants) | 29 | 14 | 20
Weeks | 64.7 [33.1 to 117] | 55.0 [20.4 to 96.1] | 78.4 [31.9 to 111]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious adverse events (SAEs) were collected from the first dose of investigational product to 30 days after the last dose of investigational product, up to approx.12 years (maximum exposure to Lapatinib (615 weeks) plus 30 days.
Description: AEs and SAEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of investigational product, according to the actual treatment received.
Groups:
- Cohort 1: Paclitaxel 80mg/Trastuzumab 4 mg/Lapatinib 1000mg: Participants received an intravenous (IV) infusion of paclitaxel 80 milligrams per meter squared (mg/m^2) over 60 minutes weekly for 3 weeks of a 4-week cycle plus an IV infusion of trastuzumab 4 mg per kilogram (mg/kg) loading dose and 2 mg/kg weekly plus a daily dose of 4 tablets of lapatinib (1000 mg) at approximately the same time every day, either 1 hour (or more) before a meal or 1 hour (or more) after a meal.
Arm/Group | Cohort 1: Paclitaxel 80mg/Trastuzumab 4 mg/Lapatinib 1000mg | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 14/29 | 6/14 | 5/20
Other Adverse Events (participants affected / at risk) | 29/29 | 13/14 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Paclitaxel 80mg/Trastuzumab 4 mg/Lapatinib 1000mg (N=29) | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg (N=14) | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg (N=20)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Cellulitis streptococcal (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Paclitaxel 80mg/Trastuzumab 4 mg/Lapatinib 1000mg (N=29) | Cohort 2: Paclitaxel 70 mg/Trastuzumab 4 mg/Lapatinib 1000 mg (N=14) | Cohort 3: Paclitaxel 80 mg/Trastuzumab 4 mg/Lapatinib 750 mg (N=20)
Anaemia (Blood and lymphatic system disorders) | 11 | 2 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Eye irritation (Eye disorders) | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 3 | 0 | 2
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 2 | 1 | 1
Visual impairment (Eye disorders) | 3 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 28 | 13 | 15
Dyspepsia (Gastrointestinal disorders) | 7 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 11 | 13
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 3 | 6
Toothache (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 17 | 6 | 4
Asthenia (General disorders) | 1 | 1 | 1
Chest pain (General disorders) | 2 | 1 | 0
Chills (General disorders) | 4 | 1 | 0
Fatigue (General disorders) | 21 | 12 | 13
Mucosal inflammation (General disorders) | 8 | 6 | 2
Non-cardiac chest pain (General disorders) | 0 | 4 | 2
Oedema peripheral (General disorders) | 5 | 4 | 0
Pain (General disorders) | 4 | 3 | 4
Peripheral swelling (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 6 | 5 | 5
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 3 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1
Candida infection (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 3 | 1 | 1
Ear infection (Infections and infestations) | 2 | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 3 | 1 | 1
Laryngitis (Infections and infestations) | 2 | 0 | 0
Localised infection (Infections and infestations) | 5 | 1 | 0
Nail infection (Infections and infestations) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Paronychia (Infections and infestations) | 2 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 3 | 1
Skin infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | 3
Urinary tract infection (Infections and infestations) | 5 | 3 | 2
Vaginal infection (Infections and infestations) | 3 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 1
Blood potassium decreased (Investigations) | 2 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 6 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 1
Weight decreased (Investigations) | 7 | 3 | 0
Weight increased (Investigations) | 1 | 1 | 0
White blood cell count decreased (Investigations) | 3 | 1 | 3
White blood cell count increased (Investigations) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 8 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 5
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 4
Dysgeusia (Nervous system disorders) | 3 | 1 | 2
Headache (Nervous system disorders) | 8 | 5 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 5 | 6 | 4
Paraesthesia (Nervous system disorders) | 7 | 1 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 2 | 3
Syncope (Nervous system disorders) | 1 | 1 | 0
Toxic neuropathy (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 3 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 3 | 3 | 1
Insomnia (Psychiatric disorders) | 6 | 7 | 3
Dysuria (Renal and urinary disorders) | 3 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 8 | 11
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 25 | 9 | 17
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Mastectomy (Surgical and medical procedures) | 1 | 0 | 2
Prophylaxis (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 0 | 0
Hot flush (Vascular disorders) | 5 | 2 | 3
Hypotension (Vascular disorders) | 2 | 0 | 0
Lymphoedema (Vascular disorders) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.